CLINICAL TRIAL: NCT06715852
Title: Moving on! Can a Tailored Treatment in a Primary Care Setting Reduce Symptoms, Healthcare Consumption, Sick Leave and Prevent Pain and Hypertension in Individuals With Anxiety Disorders?
Brief Title: Moving on! A Tailored Treatment in a Primary Care Setting for Individuals With Anxiety Disorders?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2024-02725-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: A clinical intervention with a matched design and parallel arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PHYSBI: 12-week physical exercise program (Experimental): An individualized 12-week training program including 3 occasions/week of moderate-high intensity. It may also contain elements of high intensity, corresponding to 3.0-8.9 metabolic equivalents (METs), Borg Rating of Perceived Exertion (RPE) 12-17 and 60-94% of maximal heart rate. The intervention includes cardiorespiratory and resistance training where two sessions per week are group-sessions and one session per week is performed individually. A study physiotherapists will design individualized exercise programs during a single one-to-one session with the patients.
  Interventions: Behavioral: PHYSBI: a 12-week physical exercise program
- Modified eHealth Lift: a digital, evidence based lifestyle-intervention for health promotion. (Experimental): A modified and digital development of the Health Lift, an evidence based lifestyle-intervention for health promotion and prevention in primary health care. This intervention will be executed together with care manager contact according to medical guidelines. The patient receives a material consisting of separate questionnaires dealing with dietary habits, smoking, alcohol habits, physical activity, stress, living conditions, waist-hip-ratio and well-being expressed as a life ladder, present and future. Results are then converted into a health profile and a counsellor indicated what could be offered individually or in groups depending on the participant's wishes. This person-centered method ia based on strengthening the individual's own chosen health promoting activities and support for participation in municipal facilities.
  Interventions: Behavioral: Modified eHealth Lift: a digital, evidence based lifestyle-intervention for health promotion.
- Care as usual (No Intervention): Care as usual for anxiety disorders at the primary care centers.

INTERVENTIONS:
Behavioral: PHYSBI: a 12-week physical exercise program — An individualized 12-week training program including 3 occasions/week of moderate-high intensity.
  Arms: PHYSBI: 12-week physical exercise program
Behavioral: Modified eHealth Lift: a digital, evidence based lifestyle-intervention for health promotion. — Through questionnaires, the patients answers questions regarding lifestyle habits and the results are converted into a health profile. A care manager will together with the patient decide appropriate health promoting activities to engage in.
  Arms: Modified eHealth Lift: a digital, evidence based lifestyle-intervention for health promotion.

SUMMARY:
The goal of this clinical study is to investigate the effects of two different interventions in patients with anxiety disorder and who seeks help at primary care centers. The participants will choose between two interventions:

1. A 12-week physical exercise program with three training sessions per week, or
2. A modified version of eHealth Lift, a digital development of the Health Lift, an evidence based lifestyle-intervention for health promotion and prevention in primary health care.

The participant will fill in self-assessment scales and questionnaires and also have BMI and blood pressure measured at the start of the study, at 12-weeks after the study start and after 1 year.

The main question the investigators aim to answer is if the interventions are better than treatment as usual for this group of patients regarding:

* symptoms of anxiety and depression
* pain
* sleep
* alcohol habits
* fatigue
* general health
* work ability/sick leave
* physical activity
* perceived quality of life
* BMI and blood pressure
* number of health care contacts
* psychopharmaceuticals and analgesics prescribed
* health literacy

DETAILED DESCRIPTION:
Every third patient in the waiting room at a Swedish primary healthcare center is seeking help for common mental disorders including anxiety (1). Anxiety disorders substantially reduce quality of life and daily functioning and are, among mental disorders, the second leading cause of years lived with disability and the sixth-leading cause of disability globally. Anxiety disorders are also associated with elevated risks of pain, cardiovascular disease (CVD) and premature mortality (2), emphasizing the importance of finding effective treatment strategies that can be addressed in primary care.

Specific research questions:

* Can a tailored treatment and secondary prevention in a primary care setting reduce symptoms of anxiety, healthcare consumption, sick leave, pain and prevent hypertension in individuals with anxiety disorders?
* Are there long-term effects at 1 year of follow-up regarding the outcome measures?
* Is the treatment/secondary preventive strategy associated with health economic benefits?

Significance and scientific novelty: Despite the high burden of anxiety, there are major knowledge gaps when it comes to secondary preventive measures. This intervention aims to reduce anxiety, improve the quality of life, work ability and health in primary health care patients with anxiety disorders. Little research has focused on lifestyle improvements or exercise specifically in the treatment of anxiety. In Sweden there are guidelines from The National Board of Health and welfare for treatment of depression with exercise, but guidelines for treatment of anxiety disorders are currently lacking. Also results from this study may extend the current understanding and practice in the field of treatment and secondary prevention of anxiety disorders within primary care.

This project aims to combine evidence-based interventions to tailor a lifestyle intervention with different steps focusing on patient control and participation since the individual chooses the intervention arm. Two evidence-based lifestyle interventions will combined and evaluated: the modified eHealth Lift/Care manager according to regional clinical guidelines and PHYSBI, a promising new strategy with an intensive training program, a new approach for treating anxiety disorders. If a simple intervention program in primary care can alleviate anxiety, improve quality of life, cognitive performance, and work ability, prevent pain and hypertension, this may have a great positive impact both at the individual level and from a societal perspective. The investigators hope to increase the availability of person-centered, evidence-based and cost-effective measures to promote both physical and mental health in patients with anxiety disorders. Moreover, the interventions are designed to easily be implemented in regular primary care activities.

Design of study: A clinical intervention with a matched design with two parallel arms and three assessment points (baseline, post-intervention and 1 year of follow-up).

Setting: Primary care centers in Region Västra Götaland (VGR), Sweden Participants: Patients aged 18-65 diagnosed with anxiety disorders attending 20 primary care centers (PCCs) within the VGR. Participants will be recruited by personnel at the PCCs (doctors, psychologists, nurses), through information material at the PCCs (posters, flyers and handouts) and by using the primary care system Medrave to identify and contact suitable patients. Eligibility criteria can be found elsewhere in the ClinicalTrials.gov protocol. Participants will sign a written informed consent and informed about the possibility to withdraw from the study at any time without disadvantages.

Matching: PCCs connected to a rehabilitation clinic will be assigned as intervention PCCs. Thsese PCCs will be matched for the following variables 1) size of the PCC, 2) socioeconomy as Care Need Index (CNI) and 3). Matching will be executed in order to identify suitable PCCs with care as usual (controls).

The intervention: The 10 PCCs allocated to intervention will offer all patients with a registered anxiety diagnosis in the PCCs electronic patient register as well as patients newly diagnosed with any of the above listed disorders to participate in an intervention program. The patient chooses the intervention arm, and the focus is on person-centredness, control, empowerment and participation.

The two intervention-options are:

1. Modified eHealth Lift, a digital development of the Health Lift, an evidence based lifestyle-intervention for health promotion and prevention in primary health care. This intervention will be executed together with care manager contact according to regional clinical guidelines.
2. The moderate-high intensity arm of PHYSBI, an individualized 12-week training program for anxiety disorders including 3 occasions/week. The moderate intensity arm of PHYSBI, which also will contain elements of high intensity, corresponds to 3.0-8.9 metabolic equivalents, Borg Rating of Perceived Exertion 12-17 and 60-94% of maximal heart rate. The intervention includes cardiorespiratory and resistance training in a group-session (3). The study physiotherapists design individualized exercise programs during a single one-to-one session with the patients.

CAU (PCCs allocated to non-intervention): At Swedish PCCs, care as usual (CAU) for patients with anxiety disorders can consist of visits to various healthcare professionals (such as physicians, nurses, psychologists, therapists, physiotherapists). The treatment should follow the regional guidelines, which are based on the national evidence-based clinical guidelines for anxiety disorders (National guidelines for care of depression and anxiety disorders, The Swedish National Board of Health and Welfare, Stockholm 2020). These guidelines include psychopedagogic support, psychotherapy (cognitive behavioural therapy (CBT) face-to-face or internet-mediated), psychopharmaceutical treatment and/or sick listing (preferably partial).

Outcome measures: Individual data on symptoms of anxiety, depression, general health, pain, sleep, fatigue, work ability, physical activity and perceived quality of life will be obtained through established self-assessment scales and collected for each intervention arm. Patients will self-report smoking, concurrent illnesses, pain, usage of prescribed drugs and physical activity using a questionnaire designed by the research team. Data will also be obtained from the healthcare database VEGA (Database for health-care consumption in VGR), the national Patient register, the regional prescribed drug register Digitalis, the national Prescribed drug register and the MiDAS database at Försäkringskassan (includes data on sick leave >14 days). Specification of outcomes can be found elsewhere in the ClinicalTrials.gov protocol.

Timeline and Workplan: During 2024 a Clinical Trial registration will be submitted. The investigators already have established contacts with gyms, the PHCRs and the Research and Development primary healthcare centres. During 2024 the collaborations with the primary healthcare organization, the PHCRs and health centres will be further established. A steering committee will be formed and the study procedures tested. During autumn 2024 the PCCs will be invited to participate. At the intervention PCCs, the recruitment of patients will be facilitated through a research nurse. At every PCC, a unique care manager manager which has been implemented at all PCCs in VGR since 2016 (4) handles the modified eHealth Lift, and the physiotherapists implement PHYSBI. The PHCRs will perform the PHYSBI arm and the involved PCCs will implement the modified eHealth Lift arm continuously during the intervention year of 2025. Study start date is anticipated to be in Jan 2025 and primary completion date in Dec 2026 (1 year of follow-up). Outcome data will be collected throughout the period 2025-2026. In 2026-2027 data will be processed, analyzed and scientific papers produced.

Data analysis and statistics: The majority of outcome variables are scale variables that may be treated as continuous variables and therefore primarily modelled using linear regression. These are scales for symptoms of anxiety, depression, pain, sleep, general health, perceived quality of life, sick leave days, number of health care contacts and number and types of psychopharmaceuticals prescribed. Data will be presented using descriptive statistics, including means and standard deviations for continuous variables, and frequencies and percentages for categorical variables Group differences by intervention status (modified eHealth Lift, PHYSBI, or CAU) will be assessed by Kruskal-Wallis test and chi-square tests, respectively. The average change in continuous outcomes will be analyzed using linear regression, with intervention as categorical predictor and baseline levels as covariates.

In the case of count data the investigators will test whether Poisson or negative binomial models are more appropriate than linear regression. The correlation of outcomes between patients from the same PCC will be modelled using a hierarchical linear model including PCC as random effect. A more detailed analysis of the longitudinal change will be based on repeated-measure models that also account for the correlations within individuals. Interaction terms for PCC status and time will test whether time trends differ by intervention status. Binary endpoints such as sick leave will be analyzed using logistic regression with adjustment for correlations as described for the linear models. All regression models will be adjusted for age, sex, as well as for variables on PCC-level such as socioeconomy, number of patients listed per PCC (size), and proportion of patients with anxiety diagnoses.

Power considerations: A power calculations has been performed based on 20 health centres distributed 50:50 i.e. 10 controls and 10 with two interventions. However, as patients are allowed to choose between the two intervention types (modified eHealth Lift or PHYSBI) the investigators will consider an unequal distribution of intervention types, e.g. 70:30 % for the modified eHealth Lift and PHYSBI. As the main outcome measures are continuous, Cohen's d = mean difference/standard deviation is considered as outcome measure, assuming small to medium effect size, i.e. d = 0.2 - 0.5 [51]. Power analysis was performed using a STATA procedure for one-way ANOVA. For a change (baseline to 3 months) effects sizes with d ≥ 0.2 and a power of ≥0.9 (significance level = 0.05) can be observed with a total of 320 individuals, distributed as 160 patients without intervention, 112 with the modified eHealth Lift, and 48 with PHYSBI. The same sample size will yield even larger statistical power if the group size for the modified eHealth Lift and PHYSBI were more alike.

Health-economic analyses: Cost-effectiveness analyses will be performed separately, comparing the two intervention arms to no CAU, including both direct (healthcare and pharmaceutical utilization) and indirect (long-term sickness and absenteeism from work) costs. Cost-effectiveness analyses will be based on the primary data collected within the project and based on a combination of primary data and secondary data from other sources for lifetime time perspectives. The long-term analyses will be performed using a health-economic simulation model projecting the outcomes and cost-effectiveness at the 1-year follow-up to a longer time period (5 years and lifelong).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of anxiety disorder (panic syndrome, 41.0; generalized anxiety, F41.1; mixed anxiety- and depression, F41.2 and F41.3; anxiety not otherwise specified, F41.9).
* Seeking care at primary care centers within the Region Västra Götaland.
* With or without ongoing treatment with psychoactive medication (antidepressants or anxiolytics).

Exclusion Criteria:

* Pregnancy
* Physical difficulties in performing a physical exercise program
* Pathological electrocardiogram
* Low BMI (under 17.5)
* Ongoing alcohol/substance abuse
* Ongoing exhaustion disorder or psychotic disorder
* Newly discovered (within 6 months) atrial fibrillation
* High suicide risk as assessed by the general practitioner
* Limited knowledge in the Swedish language.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety - BAI | At study start
  Established psychiatric self-assessment scale Beck Anxiety Inventory (BAI). BAI is organized in 21 items, with scoring from nothing (0 p), slightly (1 p), moderately (2p) and severely (3p) and total ratings range from nothing, minimal/mild (score 0-15), moderately (score 16-25) and severely (score 26-63).
Symptoms of anxiety - BAI | After 12-weeks intervention
  Established psychiatric self-assessment scale Beck Anxiety Inventory (BAI). BAI is organized in 21 items, with scoring from nothing (0 p), slightly (1 p), moderately (2p) and severely (3p) and total ratings range from nothing, minimal/mild (score 0-15), moderately (score 16-25) and severely (score 26-63).
Symptoms of anxiety - BAI | After one year follow-up
  Established psychiatric self-assessment scale Beck Anxiety Inventory (BAI). BAI is organized in 21 items, with scoring from nothing (0 p), slightly (1 p), moderately (2p) and severely (3p) and total ratings range from nothing, minimal/mild (score 0-15), moderately (score 16-25) and severely (score 26-63).
Symptoms of Generalized Anxiety Disorder - GAD-7 | At study start
  An established psychiatric self-assessment scale GAD-7 (Symptoms of Generalized Anxiety Disorder). A 7-item scale where anxiety severity is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety
Symptoms of Generalized Anxiety Disorder - GAD-7 | After 12-weeks intervention
  An established psychiatric self-assessment scale GAD-7 (Symptoms of Generalized Anxiety Disorder). A 7-item scale where anxiety severity is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety
Symptoms of Generalized Anxiety Disorder - GAD-7 | After one year follow-up
  An established psychiatric self-assessment scale GAD-7 (Symptoms of Generalized Anxiety Disorder). A 7-item scale where anxiety severity is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety
Symptoms of anxiety - HAD | At study start
  The established psychiatric self-assessment scale HAD (Hospital Anxiety and Depression Scale Symptoms of anxiety) is a scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Score 0-7 = Normal, 8-10 = Borderline abnormal and 11-21 = Abnormal (case).
Symptoms of anxiety - HAD | After 12-weeks intervention
  The established psychiatric self-assessment scale HAD (Hospital Anxiety and Depression Scale Symptoms of anxiety) is a scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Score 0-7 = Normal, 8-10 = Borderline abnormal and 11-21 = Abnormal (case).
Symptoms of anxiety - HAD | After one year follow-up
  The established psychiatric self-assessment scale HAD (Hospital Anxiety and Depression Scale Symptoms of anxiety) is a scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Score 0-7 = Normal, 8-10 = Borderline abnormal and 11-21 = Abnormal (case).
Symptoms of inner tension - MADRS-S; question 2 | At study start
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale); question 2, which asks about inner tension (a proxy for anxiety). The question is scaled from 0 to 6, with higher scores reflecting more severe symptoms.
Symptoms of inner tension - MADRS-S; question 2 | After 12-weeks intervention
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale); question 2, which asks about inner tension (a proxy for anxiety). The question is scaled from 0 to 6, with higher scores reflecting more severe symptoms.
Symptoms of inner tension - MADRS-S; question 2 | After one year follow-up
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale); question 2, which asks about inner tension (a proxy for anxiety). The question is scaled from 0 to 6, with higher scores reflecting more severe symptoms.

SECONDARY OUTCOMES:
Symptoms of depression - MADRS-S | At study start
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale) contains nine questions. The question are scaled from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60), with the following cut-offs: 0-6 indicate an absence of symptoms; 7-19 represent mild depression; 20-34 moderate; 35-60 indicate severe depression.
Symptoms of depression - MADRS-S | After 12-weeks intervention
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale) contains nine questions. The question are scaled from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60), with the following cut-offs: 0-6 indicate an absence of symptoms; 7-19 represent mild depression; 20-34 moderate; 35-60 indicate severe depression.
Symptoms of depression - MADRS-S | After one year follow-up
  The established psychiatric self-assessment scale MADRS-S (Montgomery-Åsberg Depression Rating Scale) contains nine questions. The question are scaled from 0 to 6, with higher scores reflecting more severe symptoms. Ratings can be added to form an overall score (from 0 to 60), with the following cut-offs: 0-6 indicate an absence of symptoms; 7-19 represent mild depression; 20-34 moderate; 35-60 indicate severe depression.
Symptoms of pain - PSQ | At study start
  The established self-assessment scale PSQ (Pain Sensitivity Questionnaire) with 17 items rated on a 11-point scale with 0 meaning "not painful at all" and 10 meaning "worst pain imaginable." Three items (items 5, 9, and 13) are not normally rated as painful and are not included in scoring. Two scores are obtained from the PSQ. The PSQ-total score is the average of all items, except for the three non-painful items. The PSQ-minor score is the average of items 3, 6, 7, 10, 11, 12, and 14 - items, on average, that are perceived as causing minor pain.
Symptoms of pain - PSQ | After 12-weeks intervention
  The established self-assessment scale PSQ (Pain Sensitivity Questionnaire) with 17 items rated on a 11-point scale with 0 meaning "not painful at all" and 10 meaning "worst pain imaginable." Three items (items 5, 9, and 13) are not normally rated as painful and are not included in scoring. Two scores are obtained from the PSQ. The PSQ-total score is the average of all items, except for the three non-painful items. The PSQ-minor score is the average of items 3, 6, 7, 10, 11, 12, and 14 - items, on average, that are perceived as causing minor pain.
Symptoms of pain - PSQ | After one year follow-up
  The established self-assessment scale PSQ (Pain Sensitivity Questionnaire) with 17 items rated on a 11-point scale with 0 meaning "not painful at all" and 10 meaning "worst pain imaginable." Three items (items 5, 9, and 13) are not normally rated as painful and are not included in scoring. Two scores are obtained from the PSQ. The PSQ-total score is the average of all items, except for the three non-painful items. The PSQ-minor score is the average of items 3, 6, 7, 10, 11, 12, and 14 - items, on average, that are perceived as causing minor pain.
Sleep quality - ISI | At study start
  The established self-assessment scale ISI (Insomnia Severity Index) includes 7 items where responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)."
Sleep quality - ISI | After 12-weeks intervention
  The established self-assessment scale ISI (Insomnia Severity Index) includes 7 items where responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)."
Sleep quality - ISI | After one year follow-up
  The established self-assessment scale ISI (Insomnia Severity Index) includes 7 items where responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. A total score of 0-7 indicates "no clinically significant insomnia," 8-14 means "subthreshold insomnia," 15-21 is "clinical insomnia (moderate severity)," and 22-28 means "clinical insomnia (severe)."
Alcohol habits - AUDIT | At study start
  The established self-assessment scale AUDIT (Alcohol Use Disorders Identification Test) including 10 items. Item 1-8 is scored with 0 to 4 points and item 9-10 with 0, 2 or 5 points. A total of 0-40 points can be obtained, where 0 to 7 indicates low risk, 8 to 15 indicates increasing risk, 16 to 19 indicates higher risk, and 20 or more indicates possible dependence.
Alcohol habits - AUDIT | After 12-weeks intervention
  The established self-assessment scale AUDIT (Alcohol Use Disorders Identification Test) including 10 items. Item 1-8 is scored with 0 to 4 points and item 9-10 with 0, 2 or 5 points. A total of 0-40 points can be obtained, where 0 to 7 indicates low risk, 8 to 15 indicates increasing risk, 16 to 19 indicates higher risk, and 20 or more indicates possible dependence.
Alcohol habits - AUDIT | After one year follow-up
  The established self-assessment scale AUDIT (Alcohol Use Disorders Identification Test) including 10 items. Item 1-8 is scored with 0 to 4 points and item 9-10 with 0, 2 or 5 points. A total of 0-40 points can be obtained, where 0 to 7 indicates low risk, 8 to 15 indicates increasing risk, 16 to 19 indicates higher risk, and 20 or more indicates possible dependence.
Fatigue - MFS | At study start
  The established self-assessment scale MFS (Mental Fatigue Scale) includes 14 items. A rating of 0 (no problem) corresponds to normal function and 1 (slight problem), 2 (fairly serious problem) and 3 (serious problem) indicate increasing problem with the symptom. A total score of above 10 implicates problems with mental fatigue and the person should consider the actual situation with work or social life.
Fatigue - MFS | After 12-weeks intervention
  The established self-assessment scale MFS (Mental Fatigue Scale) includes 14 items. A rating of 0 (no problem) corresponds to normal function and 1 (slight problem), 2 (fairly serious problem) and 3 (serious problem) indicate increasing problem with the symptom. A total score of above 10 implicates problems with mental fatigue and the person should consider the actual situation with work or social life.
Fatigue - MFS | After one year follow-up
  The established self-assessment scale MFS (Mental Fatigue Scale) includes 14 items. A rating of 0 (no problem) corresponds to normal function and 1 (slight problem), 2 (fairly serious problem) and 3 (serious problem) indicate increasing problem with the symptom. A total score of above 10 implicates problems with mental fatigue and the person should consider the actual situation with work or social life.
Health-related quality of life - EQ-5D | At study start
  The established self-assessment scale EQ-5D consist of both a visual analogue scale (EQ5D-VAS) and an index score. The EQ5D-VAS records subjective self-rated general well-being on a scale from 0-100, where a higher value corresponds to better health. The index score is derived from the EQ5D-3L survey, including 5 items with three levels of responses (no problems, some problems, and extreme problems).
Health-related quality of life - EQ-5D | After 12-weeks intervention
  The established self-assessment scale EQ-5D consist of both a visual analogue scale (EQ5D-VAS) and an index score. The EQ5D-VAS records subjective self-rated general well-being on a scale from 0-100, where a higher value corresponds to better health. The index score is derived from the EQ5D-3L survey, including 5 items with three levels of responses (no problems, some problems, and extreme problems).
Health-related quality of life - EQ-5D | After one year follow-up
  The established self-assessment scale EQ-5D consist of both a visual analogue scale (EQ5D-VAS) and an index score. The EQ5D-VAS records subjective self-rated general well-being on a scale from 0-100, where a higher value corresponds to better health. The index score is derived from the EQ5D-3L survey, including 5 items with three levels of responses (no problems, some problems, and extreme problems).
Work ability - C2WI | At study start
  The established self-assessment scale C2WI (Capacity to Work Index) including 12 items is an index to assess capacity to work in relation to common mental disorders. The items can be answered with six alternatives: Not at all, To a low degree, To a moderate degree, To a high degree, I do not know and Not relevant.
Work ability - C2WI | After 12-weeks intervention
  The established self-assessment scale C2WI (Capacity to Work Index) including 12 items is an index to assess capacity to work in relation to common mental disorders. The items can be answered with six alternatives: Not at all, To a low degree, To a moderate degree, To a high degree, I do not know and Not relevant.
Work ability - C2WI | After one year follow-up
  The established self-assessment scale C2WI (Capacity to Work Index) including 12 items is an index to assess capacity to work in relation to common mental disorders. The items can be answered with six alternatives: Not at all, To a low degree, To a moderate degree, To a high degree, I do not know and Not relevant.
Physical activity - IPAQ | At study start
  The short form of the established self-assessment scale IPAQ (The International Physical Activity Questionnaires) records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. Frequency and duration are collected separately for each specific type of activity. Both categorical and continuous indicators of physical activity can be obtained. The continuous indicator is presented as median minutes or median MET. Three levels of physical activity categories are recorded: Inactive, Minimally Active and Active.
Physical activity - IPAQ | After 12-weeks intervention
  The short form of the established self-assessment scale IPAQ (The International Physical Activity Questionnaires) records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. Frequency and duration are collected separately for each specific type of activity. Both categorical and continuous indicators of physical activity can be obtained. The continuous indicator is presented as median minutes or median MET. Three levels of physical activity categories are recorded: Inactive, Minimally Active and Active.
Physical activity - IPAQ | After one year follow-up
  The short form of the established self-assessment scale IPAQ (The International Physical Activity Questionnaires) records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. Frequency and duration are collected separately for each specific type of activity. Both categorical and continuous indicators of physical activity can be obtained. The continuous indicator is presented as median minutes or median MET. Three levels of physical activity categories are recorded: Inactive, Minimally Active and Active.
Body mass index - BMI | At study start
  Measured at primary care center as kg/m2
Body mass index - BMI | After 12-weeks intervention
  Measured at primary care center as kg/m2
Body mass index - BMI | After one year follow-up
  Measured at primary care center as kg/m2
Blood pressure - mmHg | At study start
  Measured at primary care center as mmHg.
Blood pressure - mmHg | After 12-weeks intervention
  Measured at primary care center as mmHg.
Blood pressure - mmHg | After one year follow-up
  Measured at primary care center as mmHg.
Health care contacts - registry data | At study start
  Number of health care contacts due to anxiety disorders obtained from registry data in the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Health care contacts - registry data | After 12-weeks intervention
  Number of health care contacts due to anxiety disorders obtained from registry data in the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Health care contacts - registry data | After one year follow-up
  Number of health care contacts due to anxiety disorders obtained from registry data in the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Prescribed medication - registry data | At study start
  Prescribed psychopharmaceuticals and analgesics, obtained from registry data in the Swedish Prescribed drug register and Digitalis register.
Prescribed medication - registry data | After 12-weeks intervention
  Prescribed psychopharmaceuticals and analgesics, obtained from registry data in the Swedish Prescribed drug register and Digitalis register.
Prescribed medication - registry data | After one year follow-up
  Prescribed psychopharmaceuticals and analgesics, obtained from registry data in the Swedish Prescribed drug register and Digitalis register.
Sick leave - registry data | At study start
  Extent of sick leave obtained from registry data in the MiDAS register at the Swedish Social Insurance Agency.
Sick leave - registry data | After 12-weeks intervention
  Extent of sick leave obtained from registry data in the MiDAS register at the Swedish Social Insurance Agency.
Sick leave - registry data | After one year follow-up
  Extent of sick leave obtained from registry data in the MiDAS register at the Swedish Social Insurance Agency.
Mental and Physical health - registry data | At study start
  Diagnoses of mental and physical health as ICD-10 codes (International Classification of Diseases ), obtained from the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Mental and Physical health - registry data | After 12-weeks intervention
  Diagnoses of mental and physical health as ICD-10 codes, obtained from the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Mental and Physical health - registry data | After one year follow-up
  Diagnoses of mental and physical health as ICD-10 codes, obtained from the Swedish National Patient register (hospital outpatient and inpatient care) and VEGA register (primary care data from Region Västra Götaland).
Sick leave and work ability - questionnaire | At study start
  Questions regarding extent of sick leave and ability to work in a questionnaire designed by the research team.
Sick leave and work ability - questionnaire | After 12-weeks intervention
  Questions regarding extent of sick leave and ability to work in a questionnaire designed by the research team.
Sick leave and work ability - questionnaire | After one year follow-up
  Questions regarding extent of sick leave and ability to work in a questionnaire designed by the research team.
Used psychopharmaceuticals - questionnaire | At study start
  Questions regarding usage of psychopharmaceuticals in a questionnaire designed by the research team.
Used psychopharmaceuticals - questionnaire | After 12-weeks intervention
  Questions regarding usage of psychopharmaceuticals in a questionnaire designed by the research team.
Used psychopharmaceuticals - questionnaire | After one year follow-up
  Questions regarding usage of psychopharmaceuticals in a questionnaire designed by the research team.
Physical activity - questionnaire | At study start
  Questions regarding physical activity in a questionnaire designed by the research team.
Physical activity - questionnaire | After 12-weeks intervention
  Questions regarding physical activity in a questionnaire designed by the research team.
Physical activity - questionnaire | After one year follow-up
  Questions regarding physical activity in a questionnaire designed by the research team.
Pain - questionnaire | At study start
  Questions regarding pain in a questionnaire designed by the research team.
Pain - questionnaire | After 12-weeks intervention
  Questions regarding pain in a questionnaire designed by the research team.
Pain - questionnaire | After one year follow-up
  Questions regarding pain in a questionnaire designed by the research team.
Health care consumption - questionnaire | At study start
  Questions regarding health care consumption due to mental illness in a questionnaire designed by the research team.
Health care consumption - questionnaire | After 12-weeks intervention
  Questions regarding health care consumption due to mental illness in a questionnaire designed by the research team.
Health care consumption - questionnaire | After one year follow-up
  Questions regarding health care consumption due to mental illness in a questionnaire designed by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Åberg, PhD, MD, Principal Investigator — School of Public Health and Community Medicine, University of Gothenburg
Locations (1):
- School of Public Health and Community Medicine, Institute of Medicine, University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data generated for the current study is not publicly available for ethical reasons (in order to get ethical approval, only authorized and designated researchers can have access to individual data and are not permitted to share this data), but data on group level are available from the principal investigator on reasonable request.

REFERENCES:
- [Background] Briggs A, Sculpher M, Claxton K. Decision modelling for health economic evaluation: Oup Oxford; 2006.
- [Background] Drummond MF, Sculpher MJ, Claxton K, Stoddart GL, Torrance GW. Methods for the economic evaluation of health care programmes: Oxford university press; 2015.
- [Background] Sandheimer C, Bjorkelund C, Hensing G, Mehlig K, Hedenrud T. Implementation of a care manager organisation and its association with antidepressant medication patterns: a register-based study of primary care centres in Sweden. BMJ Open. 2021 Mar 5;11(3):e044959. doi: 10.1136/bmjopen-2020-044959. PMID 33674375
- [Background] Nyberg J, Henriksson M, Aberg ND, Wall A, Eggertsen R, Westerlund M, Danielsson L, Kuhn HG, Waern M, Aberg M. Effects of exercise on symptoms of anxiety, cognitive ability and sick leave in patients with anxiety disorders in primary care: study protocol for PHYSBI, a randomized controlled trial. BMC Psychiatry. 2019 Jun 10;19(1):172. doi: 10.1186/s12888-019-2169-5. PMID 31182054
- [Background] Batelaan NM, Seldenrijk A, Bot M, van Balkom AJ, Penninx BW. Anxiety and new onset of cardiovascular disease: critical review and meta-analysis. Br J Psychiatry. 2016 Mar;208(3):223-31. doi: 10.1192/bjp.bp.114.156554. PMID 26932485
- [Background] A N. 3.5.3 Omfattning - vad går att säga? God och nära vård - Rätt stöd till psykisk hälsa. Betänkande av utredningen Samordnad utveckling för god och nära vård. In: 2021:6 SouS, editor. Stockholm 2021: ISBN 978-91-525-0019-4; 2021. p. 164-6.
- See also: Webpage for the study (in Swedish) — https://www.gu.se/forskning/moving-on

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT06715852/Prot_SAP_000.pdf